CLINICAL TRIAL: NCT00645515
Title: Ziprasidone Versus Risperidone In The Treatment Of Chronic Schizophrenia: A Six Months, Double Blind Randomized, Parallel Group Study
Brief Title: A Study Comparing the Safety and Efficacy of Ziprasidone and Risperidone for the Treatment of Chronic Schizophrenia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated on November 20, 2003 because of poor recruitment. This study was not terminated due to safety/efficacy.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1281065
Record Dates: First submitted 2008-03-20; First posted 2008-03-27 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — ziprasidone; Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Ziprasidone
- Arm B (Active Comparator)
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Ziprasidone — Initial dose of 40 mg capsules twice daily on Days 1-3; dose could be flexibly changed within the range of 40 to 80 mg twice daily for the remainder of the study; treatment duration was 24 weeks.
  Other Names: Geodon, Zeldox
  Arms: Arm A
Drug: Risperidone — Initial dose of 10 mg once daily on Days 1-3; dose could be flexibly changed within the range of 3 to 9 mg twice daily for the remainder of the study; treatment duration was 24 weeks.
  Arms: Arm B

SUMMARY:
The purpose of this study is to compare the safety of ziprasidone and risperidone for the treatment of chronic schizophrenia. The primary purpose is to differentiate the effects of ziprasidone and risperidone on extrapyramidal side effects and the secondary purpose is to compare their tolerability and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia
* CGI-S score of 4 or less at baseline

Exclusion Criteria:

* Concurrent antipsychotic treatment
* Treatment with antidepressants or mood stabilizers within 2 weeks of randomization
* Acute exacerbation of schizophrenia within 3 months of baseline

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2003-06; Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Simpson-Angus Scale (SAS) scores at Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24 | Day 1 and Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24

SECONDARY OUTCOMES:
Change from baseline in cognitive function assessment at Weeks 4 and 24 | Day 1 and Weeks 4 and 24
Change from baseline in Patient Preference Scale (PPS) at Weeks 4, 10, 12, 16, and 24 | Day 1 and Weeks 4, 10, 12, 16, and 24
Changes in Sexual Functioning Questionnaire at Weeks 1, 4, 12, 16, and 24 | Day 1 and Weeks 1, 4, 12, 16, and 24
Change from baseline in Cuestionario Sevilla at Weeks 1, 4, 12, 16, and 24 | Day 1 and Weeks 1, 4, 12, 16, and 24
Change from baseline in Modified Resource Utilization Questionnaire (RUQ) scores at Weeks 3, 4, 6, 10, 12, 16, and 24 | Day 1 and Weeks 3, 4, 6, 10, 12, 16, and 24
Laboratory tests and electrocardiogram at Week 24 | Screening and Week 24
Adverse events on Day 1 and Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24 | Day 1 and Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24
Change from baseline in Clinical Global Impressions-Severity (CGI-S) scale scores at Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24 | Day 1 and Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24
Clinical Global Impressions-Improvement (CGI-I) scale scores at Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24 | Day 1 and Weeks 1, 2, 3, 4, 6, 10, 12, 16, and 24
Change from baseline in Positive and Negative Syndrome Scale (PANSS) total scores and negative subscale scores at Weeks 4, 10, 12, 16, and 24 | Day 1 and Weeks 4, 10, 12, 16, and 24
Barnes Akathisia Scale (BAS) and Abnormal Involuntary Movements Scale (AIMS) scores at Weeks 4, 10, 12, 16, and 24 | Day 1 and Weeks 4, 10, 12, 16, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Spain (3):
  - Pfizer Investigational Site, Bilbao, Vizcaya
  - Pfizer Investigational Site, Getxo, Vizcaya
  - Pfizer Investigational Site, Madrid

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1281065&StudyName=A%20study%20comparing%20the%20safety%20and%20efficacy%20of%20ziprasidone%20and%20risperidone%20for%20the%20treatment%20of%20chronic%20schizophrenia